CLINICAL TRIAL: NCT05915702
Title: A Multicenter, Randomized, Prospective Double-blind, Cross-over Phase 3 Study to Evaluate the Efficacy and Safety of 0.04 mmol Gd/kg Body Weight of Gadoquatrane for MRI in Adults With Known or Suspected Pathology of the Central Nervous System (CNS), Compared to 0.1 mmol Gd/kg Approved Macrocyclic Gadolinium-based Contrast Agents (GBCAs)
Brief Title: A Study to Compare How Well Gadoquatrane Works and Its Safety With an Already Available Contrast Agent for MRI in People With Known or Suspected Brain or Spinal Cord-related Problems
Acronym: Quanti CNS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 21181; 2022-501884-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging; Central Nervous System Pathology
MeSH Terms: interventions — gadobutrol; gadoterate meglumine; gadoteridol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The site staff in charge of the preparation and administration of study intervention will be unblinded and will not be involved in any evaluation of safety and efficacy. The site staff in charge of conducting all other study procedures as per the schedule of activities (SoA) will remain blinded to the study intervention administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gadoquatrane - Approved Macrocyclic GBCA (Experimental): Participants will receive one intravenous injection of gadoquatrane before or during MRI in Period 1, followed by one intravenous injection of any approved macrocyclic GBCA before or during MRI in Period 2.
  Interventions: Drug: Gadoquatrane (BAY1747846); Drug: Gadobutrol; Drug: Gadoterate meglumine; Drug: Gadoteridol
- Approved Macrocyclic GBCA - Gadoquatrane (Experimental): Participants will receive one intravenous injection of any approved macrocyclic GBCA before or during MRI in Period 1, followed by one intravenous injection of gadoquatrane before or during MRI in Period 2.
  Interventions: Drug: Gadoquatrane (BAY1747846); Drug: Gadobutrol; Drug: Gadoterate meglumine; Drug: Gadoteridol

INTERVENTIONS:
Drug: Gadoquatrane (BAY1747846) — 0.04 mmol Gd/kg body weight, solution for intravenous injection, single dose
Drug: Gadobutrol — Approved standard of care macrocyclic GBCA, 0.1 mmol Gd/kg body weight, solution for intravenous injection, single dose
Drug: Gadoterate meglumine — Approved standard of care macrocyclic GBCA, 0.1 mmol Gd/kg body weight, solution for intravenous injection, single dose
  Other Names: Gadoteric acid
Drug: Gadoteridol — Approved standard of care macrocyclic GBCA, 0.1 mmol Gd/kg body weight, solution for intravenous injection, single dose

SUMMARY:
Researchers are looking for a better way to help people with known or suspected brain or spinal cord-related problems scheduled for a "contrast-enhanced" Magnetic Resonance Imaging (MRI).

MRI is used by doctors to create detailed images of the inside of the body to identify health problems. Sometimes doctors need to inject a contrast agent into a patient's vein to perform a so called "contrast-enhanced" MRI (CE-MRI). Such CE-MRI examinations may support doctors to identify certain health problems or improve the evaluation.

The contrast agents commonly used in MRI are gadolinium-based contrast agents (GBCAs). GBCAs contain a "rare earth" element called gadolinium (Gd). Gadoquatrane is a new contrast agent under development with a lower amount of Gd needed per CE-MRI.

The main purpose of this study is to learn whether CE-MRI scans with gadoquatrane work better than MRI scans without the use of a contrast agent (GBCA). The researchers will compare the ability to detect brain and spinal cord-related problems in gadoquatrane-MRI scans to plain-MRI scans without the use of a contrast agent.

The participants will undergo 2 MRI scans, one with gadoquatrane and one with currently used GBCA. Both contrast agents will be injected into the vein.

Each participant will be in the study for between 6 and 42 days with up to 7 doctor visits.

At the start or during the study, the doctors and their study team will:

* take blood and urine samples
* do physical examinations
* check blood pressure and heart rate
* review the MRI scans obtained in the study and decide on the diagnosis
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be >= 18 years of age inclusive, at the time of signing the informed consent form
* Participants with a clinical indication for a contrast-enhanced MRI (including MRA), with any approved standard of care macrocyclic GBCA with proven efficacy, safety and tolerability in clinical routine CE-MRI/MRA (gadobutrol, gadoterate meglumine/ gadoteric acid or gadoteridol) that is used at the site for the indication, for a known or suspected CNS pathology
* Participants who can undergo study-related procedures, including 2 contrast-enhanced MRI examinations (one with gadoquatrane and one with a comparator macrocyclic GBCA), as per participant and Investigator's judgement
* Contraceptive use by female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of nonchildbearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method during the study intervention period (at a minimum of 24 hours after the last dose of study intervention)

Exclusion Criteria:

* Considered clinically unstable or has a concurrent/concomitant condition that may significantly alter image comparability between the 2 study MRIs or between study parameters (e.g. safety, pharmacokinetics [PK] parameters) or would not allow participation for the full planned study period, in the judgement of the investigator
* Participants presenting with severe renal insufficiency, defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2, derived from a serum or plasma creatinine sample obtained within 48 hours prior to the first contrast agent injection in the study
* Participants with acute kidney injury (i.e., acute renal failure), regardless of eGFR
* History of moderate to severe allergic-like reaction to any GBCA
* Bronchial asthma considered unstable or who have had recent modification to their medical therapy
* Receipt of any contrast agent < 72 h prior to the study MRIs or planned to receive any contrast agent during the trial until 24 h +/- 4 h after the second study MRI
* Planned or expected interventional diagnostic or therapeutic procedure (e.g. biopsy or surgery in the region of interest) or change in treatment (e.g. start of chemotherapy or antiangiogenic therapy, significant change in corticosteroids dose) that may significantly alter image comparability between the 2 MRIs or other study parameters (i.e. safety/adverse events (AEs) [e.g. confounding AEs or safety events due to surgery or chemotherapy], PK parameters), from the first study MRI up to 24 h after the second study MRI
* Has received any investigational product within 30 days, or within 5 times half-life of the investigational product, whatever is shorter, prior to or concurrent with this study
* Contraindications to the administration of macrocyclic GBCAs (depending on local product label), or history of adverse reaction to gadoquatrane
* Any contraindication to MRI examinations based on institution policy and investigator's clinical judgement (e.g. some metallic implants or active implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Visualization parameter contrast Enhancement assessed by separate blinded evaluation of unenhanced and combined pre- and post-gadoquatrane MRI, by a BICR | 1 day procedure
  Contrast Enhancement will be assessed on a 4-point scale (1/No: not enhanced, 2/Moderate: weakly enhanced, 3/Good: clearly enhanced, 4/Excellent: clearly and brightly enhanced). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging
Visualization parameter delineation assessed by separate blinded evaluation of unenhanced and combined pre- and post-gadoquatrane MRI, by a BICR | 1 day procedure
  Delineation will be assessed on a 4-point scale (1/No: no or unclear delineation, 2/Moderate: some aspects of delineation, 3/Good: almost clear but not complete, 4/Excellent: clear and complete delineation). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging
Visualization parameter morphology assessed by separate blinded evaluation of unenhanced and combined pre- and post-gadoquatrane MRI, by a BICR | 1 day procedure
  Morphology will be assessed on a 3-point scale (1/Poor: no or poorly evaluable, 2/Moderate: partially evaluable, 3/Good: sufficiently evaluable). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging

SECONDARY OUTCOMES:
Visualization parameter contrast assessed by separate blinded evaluation of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  Contrast Enhancement will be assessed on a 4-point scale (1/No: not enhanced, 2/Moderate: weakly enhanced, 3/Good: clearly enhanced, 4/Excellent: clearly and brightly enhanced). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Visualization parameter delineation assessed by separate blinded evaluation of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  Delineation will be assessed on a 4-point scale (1/No: no or unclear delineation, 2/Moderate: some aspects of delineation, 3/Good: almost clear but not complete, 4/Excellent: clear and complete delineation). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Visualization parameter morphology assessed by separate blinded evaluation of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  Morphology will be assessed on a 3-point scale (1/Poor: no or poorly evaluable, 2/Moderate: partially evaluable, 3/Good: sufficiently evaluable). BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Sensitivity for the detection of lesions of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Specificity for the detection of lesions of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
The overall diagnostic clinical value of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs | 1 day procedure
  The overall diagnostic clinical value is composed of 2 elements and based on: i.the evaluation of diagnostic descriptive imaging features adapted from radiologic reporting standards (detection/exclusion of enhancing pathology; location, extent, and pattern of enhancement) on a 5-point scale (1- no diagnostic clinical value from contrast enhancement, 2- poor diagnostic clinical value from contrast enhancement, 3- moderate diagnostic clinical value from contrast enhancement, 4- good diagnostic clinical value from contrast enhancement, 5- excellent diagnostic clinical value from contrast enhancement), by the BICR and the Investigator; ii. the evaluation of patient management based on the diagnostic reporting recommendations (i.e., likely diagnosis), by the Investigator. BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging
Sensitivity for the detection of malignant lesions of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs assessed by BICR and the investigator | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Specificity for the detection of malignant lesions of combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs assessed by BICR and the investigator | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Diagnoses from combined pre- and post- gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs by the Investigator | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Confidence in diagnosis combined pre- and post- gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs by BICR and by Investigator on 4PS | 1 day procedure
  The degree of confidence will be rated on a 4-point scale: 1 = Not confident， 2 = Somewhat confident, 3 = Confident, 4 = Very confident. BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Number of lesions seen on unenhanced MRI image set and combined pre- and post-gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Number of enhancing lesions seen on combined pre- and post- gadoquatrane MRI and combined pre- and post-comparator MRI with macrocyclic GBCAs, by a BICR | 1 day procedure
  BICR = blinded independent central read / blinded independent central readers; MRI = magnetic resonance imaging; GBCAs = gadolinium-based contrast agents
Number of participants with treatment emergent adverse events, including number of serious adverse events, after administration of gadoquatrane compared to macrocyclic GBCAs reported by the investigator | Within 24 ± 4 hours after administration of gadoquatrane or any approved macrocyclic GBCAs
  GBCAs = gadolinium-based contrast agents
Number of participants with treatment emergent adverse events, including number of serious adverse events, per intensity after administration of gadoquatrane compared to macrocyclic GBCAs reported by the investigator | Within 24 ± 4 hours after administration of gadoquatrane or any approved macrocyclic GBCAs
  GBCAs = gadolinium-based contrast agents

CONTACTS AND LOCATIONS:
Locations (78):
- United States (8):
  - Halo Diagnostics - Indian Wells, Indian Wells, California
  - University of California Irvine Med. Center / Diagnostic Radiology, Neuroradiology, Orange, California
  - Biogenix Molecular, LLC, Miami, Florida
  - Northwestern Memorial Hospital - Radiology, Chicago, Illinois
  - QUEST Research Institute | Farmington Hills, MI, Farmington Hills, Michigan
  - MU Health Care - University Hospital - Radiology, Columbia, Missouri
  - Duke University School of Medicine - Early Phase Research Unit - Neurology, Durham, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Argentina (6):
  - Fundacion Cientifica del Sur | Centro de Lomas de Zamora - Imaging Interventionism Department, Lomas de Zamora, Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming | Sede Central - Departamento de Diagnostico por Imagenes, CABA, Ciudad Auton. de Buenos Aires
  - Sanatorio Otamendi | Imaging Diagnostic Center, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Centro de Diagnostico Enrique Rossi | Departamento de Investigacion Clínica, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Sanatorio Allende | Departamento de Investigación Clínica, Córdoba
  - Clinica Universitaria Reina Fabiola | Consultorios Externos, Córdoba
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Central Onco Hospital | Independent Medical Diagnostic Laboratory Mediscan, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Georgi | Base II - Imaging Diagnostic Department, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - University Multiprofile Hospital For Active Treatment 'Alexandrovska' EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Prof. Dr. Alexander Chirkov EAD, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski | Radiology Department, Sofia
  - University Hospital for Active Treatment Tsaritsa Joanna - ISUL | Radiology Department, Sofia
  - MHAT Sveta Marina EAD, Varna
- Canada (2):
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - London Health Sciences Centre (LHSC) - University Hospital, London
- China (9):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Captial Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hosp. Sun Yat-Sen Univ., Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (6):
  - Fakultní nemocnice Brno - Klinika radiologie a nukleární medicíny, Brno, South Moravian
  - Fakultní nemocnice Ostrava, Ostrava - Poruba
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Fakultní Thomayerova nemocnice - RDG radiodiagnostické oddelení, Prague
- France (3):
  - Center Hospitalier Michallon - Grenoble, Grenoble
  - Centre Hospitalier Lyon Sud - Service d'imagerie, Pierre-Bénite
  - Centre Hospitalo-Universitaire de Strasbourg, Strasbourg
- Germany (4):
  - Uniklinik Augsburg / Radiologie, Augsburg, Bavaria
  - Universitätsklinikum Essen - Institut für Diagnostische und Interventionelle Radiologie und Neuroradiologie - 21181, Essen, North Rhine-Westphalia
  - St. Franziskus-Hospital GmbH, Münster, North Rhine-Westphalia
  - Uniklinik Kiel /Radiologie und Neuroradiologie, Kiel, Schleswig-Holstein
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont - Idegsebeszeti Klinika, Debrecen
  - Szent Damján Görögkatolikus Kórház - Neurologiai es Stroke Osztaly, Kisvárda
  - Pecsi Tudomanyegyetem Klinikai Kozpont - Idegsebeszeti Klinika, Pécs
  - Trial Pharma Kft. Szeged, Szeged
- Italy (3):
  - ASL Della Provincia Di Barletta Andria Trani_Ospedale L.Bonomo - Radiodiagnostica, Andria, Apulia
  - Azienda Ospedaliero-Universitaria Sant'Andrea - UOC Neuroradiologia, Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Radiologia diagnostica per immagini 2 Neuroradiologia, Bergamo, Lombardy
- Japan (10):
  - Kure Kyosai Hospital, Kure, Hiroshima
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - National Hospital Organization Kanazawa Medical Center | Clinical Trial Management Office, Kanazawa, Ishikawa-ken
  - Japan Organization of Occupational Health and Safety Kagawa Rosai Hospital, Marugame, Kagawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - National Hospital Organization Kanmon Medical Center, Shimonoseki, Yamaguchi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Osaka
- South Korea (3):
  - Konkuk University Medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Inje University Busan Paik Hospital, Busan
- Sweden (3):
  - Karolinska University Hospital, Huddinge Neuroradiology, Stockholm
  - Karolinska University Hospital, Solna Neuroradiology, Stockholm
  - Uppsala University Hospital, Neuroradiology Department, Uppsala
- Turkey (Türkiye) (6):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Binali Yildirim Universitesi Mengucek Gazi EAH - Radyoloji, Erzincan
  - Koc Universitesi Tip Fakultesi - Radyoloji, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - Ondokuz Mayis Uni Tip Fakultesi, Samsun
- United Kingdom (3):
  - Queen Elizabeth University Hospital, Glasgow, Glasgow City
  - Cardiff and Vale University Health Board | University Hospital of Wales - Nephrology and Transplant, Cardiff
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.